CLINICAL TRIAL: NCT05346653
Title: The Hemodynamic Effects of Sodium-Glucose Co-Transporter 2 Inhibitors (SGLT2i) in Acute Decompensated Heart Failure
Brief Title: The Hemodynamic Effects of SGLT2i in Acute Decompensated Heart Failure
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment goals were not met.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB22-0346
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Results first posted 2023-12-06 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Acute Decompensated Heart Failure
Keywords: SGLT2i

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SGLT2i (Active Comparator): Participants will be treated with a SGLT2i during their ICU stay. The SGLT2i and heart failure care will be managed according to routine care, and data will be collected from the participant's medical record.
  Interventions: Drug: SGLT2i
- No SGLT2i (Active Comparator): Participants will not be treated with a SGLT2i during their ICU stay. Heart failure care will be managed according to routine care, and data will be collected from the participant's medical record.
  Interventions: Other: No SGLT2i

INTERVENTIONS:
Drug: SGLT2i — dapagliflozin (10 mg daily)
  Arms: SGLT2i
Other: No SGLT2i — No SGLT2i
  Arms: No SGLT2i

SUMMARY:
The main purpose of this study is to observe hemodynamic effects of initiating sodium-glucose co-transporter 2 inhibitors (SGLT2i) in patients admitted to the intensive care unit (ICU) with acute decompensated heart failure.

DETAILED DESCRIPTION:
The exact mechanism of cardiovascular benefit from SGLT2i continues to be the source of further research. The investigators hypothesize that heart failure patients with acute decompensated heart failure will similarly benefit from the SGLT2i-associated natriuresis and diuresis. This mechanism should improve invasive hemodynamics during an inpatient ICU stay.

This is a prospective, randomized controlled study to assess cardiac benefit of SGLT2i in 40 consecutive patients admitted to University of Chicago Cardiac Intensive Care Unit (CCU) Advanced Heart Failure Service. Subjects will be randomized 1:1 to one of two routine care arms: treatment with an SGLT2i [dapagliflozin 10 mg daily] or no SGLT2i. After randomization, your SGLT2i and heart failure care will be managed according to routine care, and the investigators will collect the subject's medical data. The patient's treating physician will be able to override randomization assignment if they determine that the assignment is not in the patient's best interest.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Heart Failure Reduced ejection fraction (HFrEF) of 40 or less
3. Estimated glomerular filtration rate (eGFR) > 30milliliters(ml)/minute(min)/1.73 meter(m)2
4. Admitted to CCU by advanced heart failure service for decompensated heart failure requiring continuous hemodynamic monitoring with a pulmonary artery catheter

Exclusion Criteria:

1. Diagnosis of type 1 diabetes mellitus
2. eGFR < 30ml/min/1.73m2
3. age < 18 years old
4. Jehovah's witnesses
5. Diagnosis of group 1 pulmonary arterial hypertension
6. Insulin requirement above standard low dose sliding scale
7. Patients with a history of diabetic ketoacidosis (DKA)
8. Allergies to SGLT2i medications
9. History of intolerance to SGLT2i medications
10. Patients listed for cardiac transplantation or on mechanical support
11. Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Grinstein, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SGLT2i | No SGLT2i
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 1 subject consented to the study but was not randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | SGLT2i | No SGLT2i | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Change in Indirect Fick Cardiac Index
Description: Measured by pulmonary artery catheter
Time Frame: 4 days
Population: Only 1 subject consented to the study and was not eligible for randomization.
Arm/Group | SGLT2i | No SGLT2i
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Pulmonary Capillary Wedge Pressure (PCWP)
Description: Measured by pulmonary artery catheter
Time Frame: 4 days
Population: Only 1 subject consented to the study and was not eligible for randomization.
Arm/Group | SGLT2i | No SGLT2i
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Only one subject consented for the study and was not eligible to be randomized.
Arm/Group | SGLT2i | No SGLT2i
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT05346653/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/53/NCT05346653/ICF_001.pdf